CLINICAL TRIAL: NCT06445348
Title: Morphometric Analysis of Sub Axial Cervical Spine Pedicle in Egyptian Population
Brief Title: Analysis of Sub Axial Cervical Pedicle Spine Based on CT
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Michael Atef Mikhaeel, physician, Assiut University
Other Study IDs: Cervical pedicle screw
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cervical Pedicle Screw

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Cervical pedicle screw — cervical pedicle screw

SUMMARY:
The aim of study to analyze morphometry of sub axial cervical spine pedicle in an Egyptian population based on computed tomography (CT) and thus asses the safety and feasibility of cervical pedicle screw in the sub axial cervical spine

DETAILED DESCRIPTION:
Cervical pedicle screw (CPS) fixation is found to be superior compared with lateral mass screws because it provides more axial, bending and torsional stability and has a low risk of loosening with cyclical loading . Despite biomechanical superiority, CPS fixation is not universally accepted among surgeon s because their accuracy and safety remain technically challenging because of the close proximity of vital structures as spinal cord and vertebral artery and inherent variability in pedicle at each level. In addition. limited space is available for screw placement because of complex of cervical spine vertebrae. Therefore, the risk of complication due to screw violation of the adjacent vascular and neural structures is expected to be high when performing the operation without a clear understanding of morphometric characteristics of the pedicle .Morphometry of the cervical pedicles was studied before using cadavers but comparative computed tomography (CT) data from the age matched population shown significant differences. Recent advances in CT have made anatomic measurements more accurate. The present study was undertaken to determine the 3-dimensional pedicle geometry by calculating variables like pedicle length (PL). Pedicle height (PH). Pedicle width (PW), Pedicle axis length (PAL), Pedicle transverse angulation (PTA), Pedicle sagittal angulation (PSA), Superior pedicle distance (SPD), and lateral pedicle distance (LPD). Fortunately, computed tomography (CT) scanning become a routine preoperative examination in spinal surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* Individuals from 16 to 65 years old present to Assuit university hospital and undergo cervical spine CT scan for unrelated cause

Exclusion Criteria:

* individuals with a history of cervical spine abnormalities.
* individuals with previous cervical spine injury
* individuals with congenital or developmental malformations of cervical spine patients with inflammatory. infectious, neoplastic condition

Ages: 16 Years to 65 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Sample size was calculated using Epi- Info7. According to results of previous study (put ref.) , the pullout strength failed by fracture of pedicle screw in 40% of patients undergoing cervical spine CT. Based on this percentage, confidence limits of 7% and a confidence level of 80%, the sample needed for the study was estimated to be about 80 patients.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2025-05-21 (Estimated); Study Completion 2026-06-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of feasibility of sub axial cervical spine pedicle | Baseline
  Morphometric Analysis of sub axial cervical spine pedicle in Egyptian population

REFERENCES:
- [Background] Farooque K, Yadav R, Chowdhury B, Gamanagatti S, Kumar A, Meena PK. Computerized Tomography-Based Morphometric Analysis of Subaxial Cervical Spine Pedicle in Asymptomatic Indian Population. Int J Spine Surg. 2018 Aug 3;12(2):112-120. doi: 10.14444/5017. eCollection 2018 Apr. PMID 30276069